CLINICAL TRIAL: NCT05394675
Title: A Phase 1, First-in-Human Study of DS-9606a in Patients With Tumor Types Known to Express Claudin-6 (CLDN6)
Brief Title: A Study of DS-9606a in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS9606-137; 2022-000120-38 (EudraCT Number); REFMAL 823 (Other: Sarah Cannon Development Innovations, LLC])
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Cancer; Metastatic Cancer; Germ Cell Tumor
Keywords: Advanced Cancer; Metastatic Cancer; DS-9606a; Germ Cell Tumor
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation: DS-9606a (Experimental): Participants who will receive an intravenous (IV) dose of DS9606a starting at 0.016 mg/kg every 3 weeks.
  Interventions: Drug: DS-9606a

INTERVENTIONS:
Drug: DS-9606a — Intravenous infusion

SUMMARY:
This study will assess the safety and tolerability of DS-9606a in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, phase 1, dose escalation study of the anti-CLDN6 ADC, DS-9606a, given as a single agent to patients with solid tumors. The primary objectives are to investigate the safety and tolerability of DS-9606a and to determine the maximum tolerated dose (MTD) and recommended doses for expansion (RDE/RDEs) in advanced solid tumors.

The secondary objectives of the study are to assess the pharmacokinetic properties and immunogenicity of DS-9606a, investigate the objective response rate (ORR), duration of response (DOR), disease control rate (DCR), time to response (TTR) and progression free survival (PFS) of DS-9606a, according to RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old at the time of written informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Availability of archived tumor tissue samples; patients with germ cell tumors without archived tumor samples may be allowed with approval
* Has a left ventricular ejection fraction (LVEF) ≥50% as determined by either an echocardiogram (ECHO) or multigated acquisition scan (MUGA) within 28 days before the start of study treatment
* Adequate bone marrow and organ function within 7 days before the start of study treatment
* Life expectancy ≥3 months
* Adequate treatment washout period prior to start of study treatment
* Male patients with female partners of childbearing potential and female patients of child-bearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study for at least 6 months (for males) and for at least 7 months (for females) after the last dose of study drug. Males must agree not to freeze or donate sperm throughout the study period for at least 6 months after final administration of study drug. Investigators will advise male patients on the conservation of sperm prior to study treatment. Females must agree not to donate or retrieve ova for own use throughout the study period and for at least 7 months after final study drug administration.
* Histologically- or cytologically-documented locally advanced or metastatic cancers, including but not limited to: ovarian cancer (including fallopian tube and primary peritoneal carcinoma), germ cell tumors, uterine and endometrial cancers, pancreatic adenocarcinoma, non-squamous NSCLC, or gastric cancer
* Disease progression with standard of care therapies for metastatic disease known to confer benefit, or are intolerant to or refuse standard treatment.

Exclusion Criteria:

* Has history or current presence of central nervous system metastases, except for participants who have completed radiotherapy or surgery ≥4 weeks before the start of treatment, and fulfill all criteria (no evidence of disease progression in the CNS and no requirement for chronic corticosteroids) within 2 weeks before the start of treatment
* Other invasive malignancy within 2 years; prior or concurrent non-invasive malignancies and/or patients with localized malignancies that were treated with curative intent who remain disease-free and are considered low likelihood for recurrence may be enrolled
* History of myocardial infarction or unstable angina within 6 months before study treatment
* Has a history of symptomatic congestive heart failure (New York Heart Association classes II-IV) or a serious cardiac arrhythmia requiring treatment
* Has a corrected QT interval by Fridericia's formula (QTcF), of >470 ms based on the average of triplicate 12-lead electrocardiogram (ECG) per local read
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Has an uncontrolled infection requiring ongoing or long-term therapy
* Has a known active hepatitis or uncontrolled hepatitis B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLT) in Participants Receiving DS-9606a | Cycle 1 Day 1 through Day 21 of Cycle 2 (each cycle is 21 days)
Number of Participants with Treatment-emergent Adverse Events (TEAEs) in Participants Receiving DS-9606a | Cycle 1 Day 1 to 90 days after last dose, up to 42 months (each cycle is 21 days)

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve (AUC) | Cycles 1-5, Day 1:pre-dose, end of flush, 4 hrs & 8 hrs post-dose (Cycles 1,3, &5 only); Cycle 1 & 3,Day 2; Cycle 1 & 3,Days 4,8, & 15; Cycle 2,Days 8 & 15;Cycle 4 & 6, & up to Cycle 10,Day 1 & pre-dose every cycle, up to 42 months (each cycle = 21 days)
Pharmacokinetic Parameter Maximum Concentration (Cmax) | Cycles 1-5, Day 1:pre-dose, end of flush, 4 hrs & 8 hrs post-dose (Cycles 1,3, &5 only); Cycle 1 & 3,Day 2; Cycle 1 & 3,Days 4,8, & 15; Cycle 2,Days 8 & 15;Cycle 4 & 6, & up to Cycle 10,Day 1 & pre-dose every cycle, up to 42 months (each cycle = 21 days)
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) | Cycles 1-5, Day 1:pre-dose, end of flush, 4 hrs & 8 hrs post-dose (Cycles 1,3, &5 only); Cycle 1 & 3,Day 2; Cycle 1 & 3,Days 4,8, & 15; Cycle 2,Days 8 & 15;Cycle 4 & 6, & up to Cycle 10,Day 1 & pre-dose every cycle, up to 42 months (each cycle = 21 days)
Pharmacokinetic Parameter Trough Concentration (Ctrough) | Cycles 1-5, Day 1:pre-dose, end of flush, 4 hrs & 8 hrs post-dose (Cycles 1,3, &5 only); Cycle 1 & 3,Day 2; Cycle 1 & 3,Days 4,8, & 15; Cycle 2,Days 8 & 15;Cycle 4 & 6, & up to Cycle 10,Day 1 & pre-dose every cycle, up to 42 months (each cycle = 21 days)
Overall Response Rate of DS-9606a as Assessed by the Investigator in Participants Receiving DS-9606a | Cycle 1 Day 1 and then every 6 weeks for 24 weeks, and then every 12 weeks, up to 42 months (each cycle is 21 days)
Duration of Response (DoR) as Assessed by the Investigator in Participants Receiving DS-9606a | Cycle 1 Day 1 and then every 6 weeks for 24 weeks, and then every 12 weeks, up to 42 months (each cycle is 21 days)
Disease Control Rate (DCR) as Assessed by the Investigator in Participants Receiving DS-9606a | Cycle 1 Day 1 and then every 6 weeks for 24 weeks, and then every 12 weeks, up to 42 months (each cycle is 21 days)
Time to Response (TTR) as Assessed by the Investigator in Participants Receiving DS-9606a | Cycle 1 Day 1 and then every 6 weeks for 24 weeks, and then every 12 weeks, up to 42 months (each cycle is 21 days)
Progression-free Survival (PFS) as Assessed by the Investigator in Participants Receiving DS-9606a | Cycle 1 Day 1 and then every 6 weeks for 24 weeks, and then every 12 weeks, up to 42 months (each cycle is 21 days)
Percentage of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) and Percentage of Participants Who Have Treatment-emergent ADA | Cycle 1 Days 1 and 15, Cycles 2 and 3 Day 1, Cycle 4 Day 1 and every 4 cycles thereafter on Day 1, up to 42 months (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Daiichi Sankyo
Locations (7):
- United States (5):
  - SCRI at HealthONE, Denver, Colorado
  - Florida Cancer Specialists & Research Institute, LLC, Fort Myers, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London
  - The Royal Marsden NHS Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/